CLINICAL TRIAL: NCT06784986
Title: Impact of Using the Airseal System with Ultra-low Pneumoperitoneum in Patients Undergoing Robot-assisted Radical Prostatectomy: a Prospective, Comparative, Randomized Clinical Study.
Acronym: ARCO2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brazilian Institute of Robotic Surgery (Other)
Collaborators: Hospital Mater Dei Salvador (Unknown)
Responsible Party: Principal Investigator, NILO JORGE CARVALHO LEÃO BARRETO, MD, Brazilian Institute of Robotic Surgery
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 82409124.1.1001.5128
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Prostate Carcinoma; Prostate Neoplasm; Pain Intensity Assessment; Quality of Life (QOL)
Keywords: pneumoperitoneum; airseal; pneumoperitoneum in prostate neoplasm
MeSH Terms: conditions — Prostatic Neoplasms; Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Insufflator and Trocar (Other): Subjects enrolled in this study arm will undergo robot-assisted radical prostatectomy using a conventional CO2 insufflation system. This system maintains standard intra-abdominal pressure (12-15 mmHg) and is widely used in clinical practice.
  Interventions: Device: The Conventional Insufflation System
- AirSeal® System-Interventional (Experimental): Subjects enrolled in this study arm will undergo robot-assisted radical prostatectomy using the AirSeal® System. The device enables stable pneumoperitoneum at ultra-low pressures (6-8 mmHg), aiming to reduce complications and improve surgical outcomes.
  Interventions: Device: AirSeal® System

INTERVENTIONS:
Device: The Conventional Insufflation System — The Conventional Insufflation System employs standard CO2 insufflation techniques for maintaining intra-abdominal pressure during laparoscopic and robotic surgeries. It serves as the base for comparison with the AirSeal® System.
  Arms: Conventional Insufflator and Trocar
Device: AirSeal® System — The AirSeal® System consists of an insufflation, filtration, and recirculation system (AirSeal® IFS), a triple-lumen filtered tube set, and a valve-free trocar (AirSeal® Access Port). This innovative system allows peritoneal access and pneumoperitoneum maintenance without a mechanical seal, reducing CO2 usage and associated complications.
  Arms: AirSeal® System-Interventional

SUMMARY:
The AirSeal platform has been evaluated in urological surgeries, mainly in cases of malignant diseases 5,6. However, there is still a lack of data demonstrating the possible benefits of its use, which justifies the conduct of this research in order to aggregate such knowledge. Therefore, the objective of this prospective pilot study is to compare and evaluate the role of low-pressure pneumoperitoneum with the AirSeal system in patients with prostate cancer undergoing robot-assisted prostatectomy with those undergoing the procedure with the conventional insufflation system. We seek to provide more data on the use of AirSeal, which is associated with shorter operative times, shorter hospital stays and a lower probability of complications. In addition, we aim to ratify the effectiveness and cost-benefit of using the AirSeal system.

DETAILED DESCRIPTION:
In the last decade, robot-assisted surgery has become one of the most popular surgical approaches worldwide. This minimally invasive surgery has gained notoriety mainly for reducing surgical time, having lower amounts of bleeding, among other benefits, resulting in fewer postoperative complications. However, patients with neoplasia usually have several comorbidities, and lower intra-abdominal pressure (IAP) during surgery is essential.

High-pressure pneumoperitoneum allows for a satisfactory working space and ideal visualization of the surgical field, shortening operative time and blood loss and, ultimately, improving surgical performance. On the other hand, however, several complications are related to the use of CO2, mainly in patients with compromised pulmonary and cardiac function. Innovative valveless low-pressure trocars, such as the AirSeal ® system (AirSeal®, ConMed, Utica, NY, USA), have been introduced and appear to be a valid alternative to the standard insufflation system based on preliminary studies. This system provides a more stable pneumoperitoneum, responding to minor changes in IAP, and is associated with a reduced rate of CO2 use, absorption, and elimination. Furthermore, CO2 use has been shown to be significantly reduced with this system, resulting in a potential reduction in CO2-related complications; this is particularly beneficial for patients with impaired cardiopulmonary function.

The AirSeal® platform has been evaluated in urological surgeries, mainly in cases of malignant disease. However, data demonstrating the potential benefits of its use are still lacking, which justifies the conduct of this research in order to add to this knowledge.

Therefore, the objective of this prospective pilot study is to compare and evaluate the role of low-pressure pneumoperitoneum with the AirSeal system in prostate cancer patients undergoing robot-assisted prostatectomy with those undergoing the procedure with the conventional insufflation system. We seek to provide more data on the use of AirSeal, which is associated with shorter operative times, shorter hospital stays and a lower probability of complications. In addition, we aim to confirm the effectiveness and cost-benefit of using the AirSeal® system.

OBJECTIVES The objective is to compare intraoperative and postoperative complications in patients undergoing robot-assisted radical prostatectomy using AirSeal versus those who did not use AirSeal.

METHODOLOGY This is a prospective, randomized study with two comparative arms, whose subjects will undergo the procedures in a private institution in Salvador Bahia. It should last 1 year, with the start scheduled for June/2024. The population evaluated will be patients with prostate cancer who are scheduled for robotic-assisted prostatectomy to be performed by the team in question. All patients will be invited to participate in the study by signing the ICF. After signing, patients will be randomized to one of the two groups with a ratio of 1:1. The method chosen for this purpose will be randomization performed through sequential numbers kept in opaque, non-translucent and sealed envelopes, later drawn for random allocation into the groups. Randomization will be performed by the study coordinator. Randomization will be performed without the applicators of the postoperative scales knowing to which group the patients were allocated. According to the randomization, patients will be allocated to one of two groups: Group I (control): standard treatment and Group II (intervention): use of AirSeal.

A literature review will be conducted on the subject in question, seeking to add knowledge to this work. Perioperative outcomes will be compared between those who used AirSeal and those who used the standard insufflation system.

Data will be collected through patient records, in an electronic form and among the existing variables, we will address: console time; amount of blood loss; intra-abdominal pressure used and surgical complications. As well as postoperative complications: length of hospital stay; existence of paralytic ileus, pain complaints and postoperative complications. For all patients in both groups, pain levels will be measured using the verbal numeric scale (VNS) of pain in the immediate postoperative period (during post-anesthetic recovery) and then every 6 hours during the first 48 hours. The McGill Pain Questionnaire and the medication use questionnaire included in the protocol will also be administered once a week for the two weeks following the surgical procedure. In addition, the total use of opioids in both groups in the first 48 hours and in the two weeks following the procedure should be recorded. In addition, any complications and adverse effects of analgesia will be recorded. The EORTC QLQ-C30 questionnaire will be administered one week after surgery and data on postoperative ambulation will be assessed. All patients in both groups will receive a standard prescription for postoperative pain treatment according to the World Health Organization's analgesic pain scale. During hospitalization, all patients will be prescribed a mandatory systematic prescription of Dipyrone 1 gram every 6 hours intravenously. For patients allergic to Dipyrone, it should be replaced by Paracetamol 750mg every 6 hours orally. Other medications should be prescribed according to the level on the pain scale: if the pain is between 1 and 3, add Parecoxib 40 mg 24/24h to the prescription; if the pain is between 4 and 6, administer Tramadol 100 mg intravenously up to 6/6 hours; and if the pain is greater than or equal to 7, administer Morphine 2 mg 4/4 hours. At the time of hospital discharge, the patient should receive a prescription for home use of the simple analgesic that was used during hospitalization (dipyrone or paracetamol) if the pain is mild, and Tramadol 50 mg orally up to 6/6h for use if the pain is moderate or severe.

It is known that the use of opioids during surgery may also influence the control of postoperative pain, and with this in mind, there will be a standard protocol for the anesthetic procedure with standardization of medications used and their use according to the patient's weight and age.

Patients may request to be withdrawn from the study at any time. And participants will be screened according to the inclusion and exclusion criteria described below.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prostate cancer who will undergo robotic prostatectomy;

Exclusion Criteria:

* Patients over 65 and under 18 years of age;
* Patients allergic to NSAIDs and/or Morphine and/or Tramadol;
* Patients with chronic renal failure;
* Patients with recurrence, metastasis and other existing neoplasms.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Variance in Intra-abdominal Pressure with the AirSeal System | Day 1 (Day of Procedure)
  The primary aim of this study is to compare the variance in intra-abdominal pressure (IAP) during robotic-assisted radical prostatectomy between patients using the AirSeal System and those using a conventional CO2 insufflation system. The AirSeal System is expected to provide a more stable IAP at ultra-low pressures (6-8 mmHg) compared to the standard pressures (12-15 mmHg) maintained by the conventional insufflator.

SECONDARY OUTCOMES:
Reduction in Blood Loss with the AirSeal System | Day 1 (Day of Procedure)
  This study will measure the total blood loss during the surgical procedure in patients using the AirSeal System versus those using the conventional insufflation system. Lower blood loss is hypothesized with the AirSeal System due to better surgical visibility and lower pressure variability.
Length of Hospital Stay | Duration of hospital stay (up to 7 days)
  The length of hospital stay will be recorded for all participants. Patients using the AirSeal System are expected to have a shorter hospital stay due to reduced complications and better recovery.
Incidence of Postoperative Complications | Up to 2 weeks post-procedure
  Postoperative complications, including paralytic ileus, respiratory issues, and other adverse events, will be compared between the two groups. The AirSeal System is hypothesized to lower the incidence of these complications.

CONTACTS AND LOCATIONS:
Overall Officials: NILO J. MD, Principal Investigator — Brazilian Institute of Robotic Surgery
Locations (2):
- Brazil (2):
  - Instituto Brasileiro de Cirurgia Robotica, Salvador, Estado de Bahia
  - Hospital Mater Dei Salvador, Salvador, Estado de Bahia

REFERENCES:
- [Background] Razdan S, Ucpinar B, Okhawere KE, Badani KK. The Role of AirSeal in Robotic Urologic Surgery: A Systematic Review. J Laparoendosc Adv Surg Tech A. 2023 Jan;33(1):21-31. doi: 10.1089/lap.2022.0153. Epub 2022 Jun 7. PMID 35671523
- [Background] Horstmann M, Horton K, Kurz M, Padevit C, John H. Prospective comparison between the AirSeal(R) System valve-less Trocar and a standard Versaport Plus V2 Trocar in robotic-assisted radical prostatectomy. J Endourol. 2013 May;27(5):579-82. doi: 10.1089/end.2012.0632. Epub 2013 Feb 5. PMID 23186377
- [Background] Feng TS, Heulitt G, Islam A, Porter JR. Comparison of valve-less and standard insufflation on pneumoperitoneum-related complications in robotic partial nephrectomy: a prospective randomized trial. J Robot Surg. 2021 Jun;15(3):381-388. doi: 10.1007/s11701-020-01117-z. Epub 2020 Jul 6. PMID 32632561
- [Background] Bhat KRS, Raghunath SK, Srivatsa N, Tejus C, Vishruth K, Kumar RA. Outcomes of Minimally Invasive Radical Prostatectomy-a Contemporary Review. Indian J Surg Oncol. 2020 Dec;11(4):580-588. doi: 10.1007/s13193-020-01125-3. Epub 2020 Jun 11. PMID 33299276
- [Background] Balayssac D, Selvy M, Martelin A, Giroudon C, Cabelguenne D, Armoiry X. Clinical and Organizational Impact of the AIRSEAL(R) Insufflation System During Laparoscopic Surgery: A Systematic Review. World J Surg. 2021 Mar;45(3):705-718. doi: 10.1007/s00268-020-05869-5. Epub 2020 Nov 30. PMID 33258023